CLINICAL TRIAL: NCT02662738
Title: The Effect of a Natural Extract on Glucose Fluxes After Consumption of a Wheat Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FDS-NAA-1650
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Blood glucose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A wheat product (Active Comparator): A wheat product (containing 2% 13C-universally-labeled wheat) with natural fruit extract added.
  Interventions: Dietary Supplement: Natural fruit extract
- Control (Placebo Comparator): A wheat product (containing 2% 13C-universally-labeled wheat) without natural fruit extract added.
  Interventions: Other: Placebo
- Glucose solution (Other): A solution of 50g glucose of which 2% 13C-universally-labeled glucose (2%) and unlabeled glucose (98%) in 250 mL water.
  Interventions: Other: Glucose solution

INTERVENTIONS:
Dietary Supplement: Natural fruit extract
  Arms: A wheat product
Other: Placebo
  Arms: Control
Other: Glucose solution
  Arms: Glucose solution

SUMMARY:
This study is to quantify the effect of a natural fruit extract added to a wheat product on the time needed to absorb 50% of the apparent total of available exogenous carbohydrate (RaE * Time). In addition the different glucose fluxes will be quantified (RaE, EGP and GCR)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male.
* Body mass index (BMI) ≥ 18.0 and ≤ 25.0 kg/m2.
* Apparently healthy: no medical conditions which might affect the study measurements including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery and inflammatory diseases.
* Fasting blood glucose value of volunteer is ≥ 3.4 and ≤ 6.1 mmol/liter (i.e. 62- 110 mg/dl) at screening.
* HbA1c ≤ 6.5 % (48 mmol/mol).

Exclusion Criteria:

* Use of antibiotics within 3 months before Day 1; use of any other medication except paracetamol within 14 days before Day 1.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
13C (13 carbon) and D-[6,6-2H2] glucose | 0-6 hours

SECONDARY OUTCOMES:
Total blood glucose (BG) | 0-2 hours and 0-4 hours
Insulin | 0-2 hours and 0-4 hours
Endogenous glucose production (EGP) | 0-2 hours and 0-4 hours
Glucose clearance rate (GCR) | 0-2 hours and 0-4 hours
13C Metabolites of glucose (metabolomics) | 0-2 hours and 0-4 hours
12C Metabolites of glucose (metabolomics) | 0-2 hours and 0-4 hours
Postprandial hormones (Gastric inhibitory polypeptide, glucagon-like peptide-1 and Glucagon) | 0-2 hours and 0-4 hours
Selected anti-oxidants (vitamin E (alpha-tocopherol), lycopene, retinol, alpha-carotene and beta-carotene) | -5, 60, 120, 180, 240 and 300 minutes
Haematocrit | -5, 60, 120, 180, 240 and 300 minutes
Concentration of key active in extract | -5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 and 360 minutes
13CO2 in breath | 30, 30, 60, 90,120, 150, 180 and every 30 minutes up to 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tjeerd Mensinga, MD, PhD, Principal Investigator — QPS Netherlands
Locations (1):
- QPS, Groningen, Hanzeplein 1, Netherlands